CLINICAL TRIAL: NCT03291132
Title: Evaluation Study on Smoke-free Teens Programme
Brief Title: Smoke-free Teens Programme
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. LI William Ho Cheung, Associate Professor, The University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Purpose: Health Services Research
Other Study IDs: UW 15-402
Record Dates: First submitted 2017-08-17; First posted 2017-09-25 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-04

CONDITIONS: Smoking Cessation
Keywords: Smoke-free; Teens
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- training camp (Other): The Smoke-free teens will join a "2-Day-1-Night" training camp in July or August. The camp will cover a wide range of indoor, outdoor, adventure-based, experiential learning activities. Besides, the teens will be equipped with the knowledge on smoking hazards, tobacco control and smoking cessation. The teens will be taught how to deliver a brief smoking cessation intervention using the "AWARD" Model: By the end of the training camp, the teens should be confident and competent in delivering the brief smoking cessation intervention to smokers. The teens will then break down into groups to organize smoke-free programmes in their schools or in the community.
  All Smoke-free Teens will be invited to respond to the structured questionnaire at baseline (T1), immediately after the training camp (T2), and 3 (T3) and 6 months later (T4). Each group of teens will have to submit the written proposal and final report regarding the smoke-free programme to COSH at 3 (T3) and 6 (T4) months.
  Interventions: Other: training camp

INTERVENTIONS:
Other: training camp — The Smoke-free teens will join a "2-Day-1-Night" training camp in July or August. The camp will cover a wide range of indoor, outdoor, adventure-based, experiential learning activities. Besides, the teens will be equipped with the knowledge on smoking hazards, tobacco control and smoking cessation. The teens will be taught how to deliver a brief smoking cessation intervention using the "AWARD" Model: By the end of the training camp, the teens should be confident and competent in delivering the brief smoking cessation intervention to smokers. The teens will then break down into groups to organize smoke-free programmes in their schools or in the community.
  All Smoke-free Teens will be invited to respond to the structured questionnaire at baseline (T1), immediately after the training camp (T2), and 3 (T3) and 6 months later (T4). Each group of teens will have to submit the written proposal and final report regarding the smoke-free programme to COSH at 3 (T3) and 6 (T4) months.

SUMMARY:
This study aims to evaluate the effectiveness of the Smoke-free Teens Programme in strengthening youth's knowledge and attitude on smoking and health.

The objectives are:

i. To evaluate Smoke-free Teens' change in knowledge on smoking hazards, attitudes towards smoking, tobacco control and smoking cessation, and practices for promoting smoking prevention and cessation, ii. To evaluate the process and quality of smoke-free programmes organized by the Smoke-free Teens in their schools/community, and iii. To measure the number of people whom the Smoke-free Teens will deliver the smoke-free messages to.

DETAILED DESCRIPTION:
Participants (thereafter named Smoke-free Teens) Youth between Form 1 and 4 or aged 14 to 18 will be nominated by secondary schools, youth centres and uniform groups to participate in the Smoke-free Teens Programme .

Outcomes The primary outcomes include the change in (1) knowledge on smoking hazards, (2) attitudes towards smoking, tobacco control and smoking cessation, (3) practices for promoting smoking prevention and cessation, and (4) the Smoke-free Teens' satisfaction on the training camp.

The secondary outcomes are (1) the number of people participated in the school- or community-based smoke-free programmes organised by the Smoke-free Teens, and (2) the number of smokers advised and referred to existing smoking cessation services by the Smoke-free Teens.

The Smoke-free teens will join a "2-Day-1-Night" training camp organized by the Hong Kong Council of Smoking and Health(COSH) in July or August . The camp will cover a wide range of indoor, outdoor, adventure-based, experiential learning activities. Besides, the teens will be equipped with the knowledge on smoking hazards, tobacco control and smoking cessation. In addition, the teens will be taught how to deliver a brief smoking cessation intervention using the "AWARD" Model: 1) Ask about smoking, 2) Warn the smokers that at least half will be killed by smoking, 3) Advise to quit (reduce) as soon as possible, 4) Refer to cessation clinics or hotlines, and 5) Do it again until the smokers quit. By the end of the training camp, the teens should be confident and competent in delivering the brief smoking cessation intervention to smokers. After the training camp, the teens will then break down into groups to organize smoke-free programmes in their schools or in the community.

Survey instrument A structured questionnaire designed by the smoking cessation team, School of Nursing, the University of Hong Kong will be used to evaluate the training camp. The questionnaire covers four areas, including (1) knowledge on smoking hazards, (2) attitudes towards smoking, tobacco control and smoking cessation, (3) practices for promoting smoking prevention and cessation, and (4) self-efficacy to deliver smoking cessation advices. The items of the questionnaire have been adopted and modified from previous studies on smoking cessation, with well-established psychometric properties. A process evaluation form will also be developed by the smoking cessation team to assess how the teens satisfy with the training camp, and to determine whether the content of the training camp meets the learning needs and expectations of the teens.

To evaluate the smoke-free programmes organized after the training camp, each group of the Smoke-free Teens will be required to submit a written proposal to COSH. In addition, a final report that contains the information about the number of people reached by the programmes, publicity, and the process and outcomes of the programmes, will be submitted for review.

Data collection Data collection will be conducted by COSH. All Smoke-free Teens will be invited to respond to the structured questionnaire at baseline (T1), immediately after the training camp (T2), and 3 (T3) and 6 months later (T4). In addition, they will be asked to complete a process evaluation form immediately after the training camp (T2). Comments and suggestions provided by the teens in the process evaluation form will be taken into account for future improvement of the training camp. In addition, each group of teens will have to submit the written proposal and final report regarding the smoke-free programme to COSH at 3 (T3) and 6 (T4) months, respectively.

Statistical analysis The Statistical Package for Social Science (SPSS: Version 23; SPSS Inc., Chicago, Illinois, USA) for Windows will be employed to analyze the data. Descriptive statistics will be used to describe the demographic characteristics of the Smoke-free Teens. Paired samples t-test and McNemar's test will be conducted to assess the change in knowledge, attitudes and practices of the Smoke-free Teens regarding smoking, tobacco control and smoking cessation before and after the training camp. To evaluate the smoke-free programmes organized by the Smoke-free Teens after the training camp, descriptive statistics will be used to report the number of people reached by the programmes, publicity, and the process and outcomes of the programmes.

ELIGIBILITY:
Inclusion Criteria:

* be able to communicate with Cantonese, nominated by secondary schools, youth centres and uniform groups

Exclusion Criteria:

-

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1456 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Knowledge on smoking hazards at baseline level | Baseline
  Smoke-free Teens' knowledge on smoking hazards at baseline level will be measured by the scale called "knowledge on smoking hazards" in a self-reporting structured questionnaire.
The change in knowledge on smoking hazards | Baseline, immediately after the training camp, 3 months and 6 months
  The change in Smoke-free Teens' knowledge on smoking hazards immediately after the training camp, after 3 months, and after 6 months will be measured by the scale called "knowledge on smoking hazards" in a self-reporting structured questionnaire.
Attitudes towards smoking, tobacco control and smoking cessation at baseline level | Baseline
  Smoke-free Teens' attitudes towards smoking, tobacco control and smoking cessation at baseline level will be measured by the scale called "attitudes towards smoking, tobacco control and smoking cessation" in a self-reporting structured questionnaire.
The change in attitudes towards smoking, tobacco control and smoking cessation | Baseline, immediately after the training camp, 3 months and 6 months
  The change in Smoke-free Teens' attitudes towards smoking, tobacco control and smoking cessation immediately after the training camp, after 3 months, and after 6 months will be measured by the scale called "attitudes towards smoking, tobacco control and smoking cessation" in a self-reporting structured questionnaire.
Practices for promoting smoking prevention and cessation at baseline level | Baseline
  Smoke-free Teens' practices for promoting smoking prevention and cessation at baseline level will be measured by the scale called "practices for promoting smoking prevention and cessation" in a self-reporting structured questionnaire.
The change in practices for promoting smoking prevention and cessation | Baseline, 3 months and 6 months
  The change in Smoke-free Teens' practices for promoting smoking prevention and cessation after 3 months, and after 6 months will be measured by the scale called "practices for promoting smoking prevention and cessation" in a self-reporting structured questionnaire.
Self-efficacy to deliver smoking cessation advices at baseline level | Baseline
  Smoke-free Teens' self-efficacy to deliver smoking cessation advices at baseline level will be measured by the scale called "self-efficacy to deliver smoking cessation advices" in a self-reporting structured questionnaire.
The change in self-efficacy to deliver smoking cessation advices | Baseline, immediately after the training camp, 3 months and 6 months
  The change in Smoke-free Teens' self-efficacy to deliver smoking cessation advices immediately after the training camp, after 3 months, and after 6 months will be measured by the scale called "self-efficacy to deliver smoking cessation advices" in a self-reporting structured questionnaire.
Process evaluation of the training camp | immediately after the training camp
  Smoke-free Teens' feedback and views of the training camp will be measured immediately after the training camp by the scale called "process evaluation" in a self-reporting structured questionnaire.

SECONDARY OUTCOMES:
The number of people participated in the school- or community-based smoke-free programmes organized by the Smoke-free Teens after the training camp | 6 months
  During the training camp, smoke-free Teens will be taught how to deliver a brief smoking cessation intervention using the "AWARD" Model: 1) Ask about smoking, 2) Warn the smokers that at least half will be killed by smoking, 3) Advise to quit (reduce) as soon as possible, 4) Refer to cessation clinics or hotlines, and 5) Do it again until the smokers quit.
  After the training camp, the teens will be required to organize smoke-free programmes in their schools or communities so as to deliver brief smoking cessation intervention and to promote smoke-free messages in their schools and communities. The number of people participated in these school- or community-based smoke-free programmes will be measured by a final report submitted by the teens that indicate the relevant information.
The number of smokers advised and referred to existing smoking cessation services by Smoke-free Teens after the training camp | 6 months
  During the training camp, Smoke-free Teens will be taught how to deliver a brief smoking cessation intervention using the "AWARD" Model: 1) Ask about smoking, 2) Warn the smokers that at least half will be killed by smoking, 3) Advise to quit (reduce) as soon as possible, 4) Refer to cessation clinics or hotlines, and 5) Do it again until the smokers quit.
  After the training camp, the teens will organize smoke-free programmes in their schools or in the communities so as to deliver brief smoking cessation intervention and to promote smoke-free messages in their schools and communities. The number of smokers the teens advised and referred to existing smoking cessation services during these school- or community-based smoke-free programmes will be measured by a final report submitted by the teens that indicate the relevant information.

CONTACTS AND LOCATIONS:
Overall Officials: William LI, PhD, Principal Investigator — School of Nursing, the University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
The relevant anonymized patient level data, full dataset, technical appendix, and statistical code are available on reasonable request. The approval from the Principal Investigator for the purpose of data use is required.
Time Frame: After the project is completed and the results of the project has been published.
Access Criteria: Request could be sent to Principal Investigator (william3@hku.hk)

REFERENCES:
- [Derived] Chung OK, Li WHC, Ho KY, Kwong ACS, Lai VWY, Wang MP, Lam KKW, Lam TH, Chan SSC. A descriptive study of a Smoke-free Teens Programme to promote smoke-free culture in schools and the community in Hong Kong. BMC Public Health. 2019 Jan 7;19(1):23. doi: 10.1186/s12889-018-6318-4. PMID 30616578